CLINICAL TRIAL: NCT05802082
Title: The Effects of Preoperative Anxiety and Preemptive Analgesia on Postoperative Delirium in Adenotonsillectomy Surgery
Brief Title: Preoperative Anxiety and Preemptive Analgesia on Postoperative Delirium in Adenotonsillectomy Surgery
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, medical doctor, Zonguldak Bulent Ecevit University
Other Study IDs: 2019/10
Record Dates: First submitted 2023-01-19; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Preoperative Anxiety; Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P: n: 32patients: Group P: Patients administered iv 10mg/kg paracetamol 30 minutes before surgery
  Interventions: Other: The Modified Yale Preoperative Anxiety Scale (m-YPAS) of children
- Group K:n:32 patients: Group K: Patients administered iv 10mg/kg paracetamol 15 minutes before the end of surgery
  Interventions: Other: The Modified Yale Preoperative Anxiety Scale (m-YPAS) of children

INTERVENTIONS:
Other: The Modified Yale Preoperative Anxiety Scale (m-YPAS) of children — Postoperative 0,5,10,15,30,45,60.and 120 minutes , PAED and WBYAS values
  Other Names: Post-Anesthesia Recovery Agitation (PAED) is a self-limiting condition seen in children upon awakening from anesthesia in the first 15-20 minutes.; The Wong Baker Facial Pain Scale (WBYAS) is used to evaluate postoperative pain in children.

SUMMARY:
The effects of preoperative anxiety and preemptive analgesia on PAED in children undergoing adenotonsillectomy surgery.

DETAILED DESCRIPTION:
It is known that the frequency of postoperative delirium increases in children with preoperative anxiety.

The Modified Yale Preoperative Anxiety Inventory (m-YPAS) was developed as a tool to assess children's preoperative anxiety, and m-YPAS≥30 was considered 'anxious'.

Post-Anesthesia Recovery Agitation (PAED) is a self-limiting condition seen in children upon awakening from anesthesia in the first 15-20 minutes.

There are factors such as inhalation agents, preoperative anxiety and postoperative pain in its etiology.

ELIGIBILITY:
Inclusion Criteria:

* 2-10 years old,
* ASA I-II risk group
* Those who will be operated under general anesthesia under elective conditions.
* Will undergo surgery for adenoidectomy and/or tonsillectomy
* Patients whose informed consent form was read to their parents and their consent was obtained

Exclusion Criteria:

* Those whose families do not want to participate in the study,
* ASA III -IV-V patients
* Having a history of drug allergy and drug interaction,
* Having a history of systemic disease such as heart, kidney, liver failure,
* Having a history of bleeding diathesis,
* Difficult intubation expected,
* Obese,
* Emergency patients,
* Mental-motor retarded,
* Having psychiatric and neurological diseases,
* Those with chronic drug use

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 64
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Preoperative Anxiety on Postoperative Delirium in Adenotonsillectomy Surgery | During the first 2 hours postoperatively
  The relationship between the mYPAS values of the groups and the PAED scores and Wong Baker Facial Pain Scale values
Preemptive analgesia on Postoperative Delirium in Adenotonsillectomy Surgery | During the first 2 hours postoperatively
  The relationship between the mYPAS values of the groups and the PAED scores and Wong Baker Facial Pain Scale values

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided